CLINICAL TRIAL: NCT04731285
Title: Accuracy of RuiXin-FFR by Comparing With Pressure-wire-based FFR in Detecting Hemodynamically Significant Stenosis: A Prospective Multicenter Study
Brief Title: Evaluation of Accuracy of CFD-based RuiXin-FFR by Comparing With Pressure-wire-based FFR
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor, Beijing Anzhen Hospital
Other Study IDs: 201901RX
Record Dates: First submitted 2020-10-07; First posted 2021-01-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Myocardial Fractional Flow Reserve
Keywords: Coronary Artery Disease; Myocardial Ischemia; FFR; FFRCT
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pressure wire based FFR: Pressure wire based FFR was reference group
  Interventions: Diagnostic Test: Pressure wire fractional flow reserve
- CT-FFR: CFD-based RuiXin-FFR was test group
  Interventions: Diagnostic Test: CFD-based RuiXin-FFR

INTERVENTIONS:
Diagnostic Test: Pressure wire fractional flow reserve — Pressure wire is inserted into coronary arteries. The ratio of the average distal pressure and average aorta pressure is FFR.
  Groups: Pressure wire based FFR
Diagnostic Test: CFD-based RuiXin-FFR — CT-FFR was evaluated in a blinded fashion with a "Coarse-to-Fine Subpixel" algorithm for lumen contour
  Groups: CT-FFR

SUMMARY:
Coronary Artery Disease (CAD) is the top killer nowadays. Pressure-wire-based Fractional Flow Reserve (FFR) is the gold standard for measuring ischemia in coronary arteries. CFD-based RuiXin-FFR, which is noninvasive, is developed recently. But its accuracy is not verified. This is a multi-center and prospective study to evaluate the sensitivity, specificity, and accuracy of CFD-based RuiXin-FFR compared with wire-based FFR.

DETAILED DESCRIPTION:
The participants are entered with suspended CAD and angiography ischemia between 30%-90% from 6 hospitals in China. Pressure-wire-based FFR is conducted in the standard protocol by each hospital. FFR>0.8 is chosen as the threshold to indicate non-ischemia. CFD-based RuiXin-FFR is performed by Raysight Medical (Shenzhen, China). CT images are acquired in a standard protocol by each hospital. Images with poor quality are excluded in this trial. Based on these images, RuiXin-FFR reconstructs the 3D model of coronary trees and obtains RuiXin-FFR values by conducting CFD simulations in a blinded fashion. RuiXin-FFR>0.8 is chosen as the threshold to indicate non-ischemia as well. By comparing the clinical diagnosis outcome of pressure-wire-based FFR and CFD-based RuiXin-FFR, the sensitivity and specificity of the RuiXin-FFR are obtained, which is the primary end point of this trial. The secondary end point includes the measurement of accuracy, NPV, PPV and ROC of the RuiXin-FFR.

ELIGIBILITY:
Inclusion Criteria:

* able to understand the purpose of the study and sign the informed consent
* with diagnosed or confirmed coronary artery disease according to the comprehensive clinical assessment
* with CTA image indicating that the diameter of the reference vessel in the stenosis segment was ≥2mm
* with CTA image indicating that the stenosis degree of coronary artery lumen diameter ≥30% and ≤90%

Exclusion Criteria:

* prior coronary artery bypass bypass (CABG) surgery, coronary interventional therapy (PCI), artificial heart valve implantation, cardiac pacemaker or implantable defibrillator implantation
* persistent or active symptoms of clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure status (systolic pressure less than 90 mmHg), severe congestive heart failure (NYHA grade III or IV), or acute pulmonary edema
* acute myocardial infarction occurred within 7 days before inclusion
* complex congenital heart disease, sick sinus syndrome, long QT syndrome, severe arrhythmia, tachycardia, severe asthma, severe or very severe chronic obstructive pulmonary disease (COPD) and chronic renal damage (serum creatinine value > 1.5 mg/dl or creatinine clearance < 45 ml/Kg*1.73 m2)
* there are contraindications for the use of adenosine disodium triphosphate
* allergic to iodized contrast media
* pregnancy or pregnancy status unknown
* life expectancy less than 2 months
* there are any factors that other researchers consider not suitable for inclusion or completion of this study
* obvious mismatch of coronary artery CTA images
* CTA image showing calcification occupies the cross-sectional area of the lumen > 80%
* CT value standard deviation of aortic root image >30HU
* coronary artery occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised 330 stable patients with suspected or known CAD who underwent CCTA, and were referred to ICA, and FFR
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 9 days
  By comparing with pressure-wire-based FFR, the sensitivity and specificity of CFD-based RuiXin-FFR are measured

CONTACTS AND LOCATIONS:
Overall Officials: Zhanquan Li, MD, Principal Investigator — Liaoning Provincial People's Hospital
Locations (1):
- Shaoping Nie, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng Y, Wang X, Tang Z, Li T, Jiang X, Ji F, Zhou Y, Ge J, Li Z, Zhao Y, Ma C, Mintz GS, Nie S. Diagnostic accuracy of CT-FFR with a new coarse-to-fine subpixel algorithm in detecting lesion-specific ischemia: a prospective multicenter study. Rev Esp Cardiol (Engl Ed). 2024 Feb;77(2):129-137. doi: 10.1016/j.rec.2023.05.008. Epub 2023 Jul 13. English, Spanish. PMID 37453536